CLINICAL TRIAL: NCT05806346
Title: Tranexamic Acid Administration Strategies in Cardiovascular Surgery: Goal-directed Tranexamic Acid Administration Based on Viscoelastic Test vs. Empirical Tranexamic Acid Administration
Brief Title: Goal-directed vs. Empirical Tranexamic Acid Administrationin Cardiovascular Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); Helptrial (Unknown); Asan Medical Center (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: HI22C1952-1-3
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Heart Diseases; Vascular Diseases; Transfusion Related Complication; Coagulation Disorder, Blood; Fibrinolysis; Hemorrhage
MeSH Terms: conditions — Heart Diseases; Vascular Diseases; Blood Coagulation Disorders; Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: randomized prospective double-blind placebo-controlled multicenter non-inferior
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Empirical 1: TXA and Placebo administration (Active Comparator): Tranexamic acid administration, regardless of the result of rotational thromboelastometry.
  Placebo administration, at LI60 < 85 % or A10< 40 mm in EXTEM of rotational thromboelastometry
  Interventions: Drug: TXA administration; Drug: Placebo administration
- Empirical 2: TXA administration (Active Comparator): Tranexamic acid administration, regardless of the result of rotational thromboelastometry.
  Placebo discard, at LI60 ≥ 85% or A10 ≥ 40 mm in EXTEM of rotational thromboelastometry
  Interventions: Drug: TXA administration
- Goal-directed 1: Placebo administration (Experimental): Placebo administration, regardless of the result of rotational thromboelastometry.
  Tranexamic acid administration at LI60 < 85 % or A10 < 40 mm in EXTEM of rotational thromboelastometry
  Interventions: Drug: TXA administration; Drug: Placebo administration
- Goal-directed 2: TXA and Placebo administration (Experimental): Placebo administration, regardless of the result of rotational thromboelastometry.
  Tranexamic acid discard at LI60 ≥ 85% or A10 ≥ 40 mm in EXTEM of rotational thromboelastometry
  Interventions: Drug: Placebo administration

INTERVENTIONS:
Drug: TXA administration — Tranexamic acid intravenous administration
  Other Names: Tranexamic acid
  Arms: Empirical 1: TXA and Placebo administration; Empirical 2: TXA administration; Goal-directed 1: Placebo administration
Drug: Placebo administration — Placebo (normal saline) intravenous administration
  Other Names: Placebo (normal saline)
  Arms: Empirical 1: TXA and Placebo administration; Goal-directed 1: Placebo administration; Goal-directed 2: TXA and Placebo administration

SUMMARY:
The present study is a multi-center randomized prospective placebo-controlled non-inferiority trial.

The study's primary objective is to compare the amounts of postoperative bleeding using two different TXA administration strategies: empirical TXA administration vs. viscoelastic test-based goal-directed TXA administration in cardiovascular surgery.

The secondary objectives include comparing the incidents of hyper-fibrinolysis, thromboembolic complications, and postoperative seizures.

Researchers assumed that goal-directed tranexamic acid (TXA) administration using viscoelastic field tests would not be inferior to the empirical TXA administration strategy in reducing postoperative bleeding and hyper-fibrinolysis. It also would be beneficial in lowering TXA-induced thromboembolic complications and seizures.

DETAILED DESCRIPTION:
The present study is a multi-center randomized prospective placebo-controlled non-inferiority trial.

This study's primary objective is to compare the amounts of postoperative bleeding during postoperative 24 hours through chest tube drainage using two different tranexamic acid (TXA) administration strategies: empirical TXA administration vs. viscoelastic test-based goal-directed TXA administration in cardiovascular surgery.

The secondary objectives include determining the inter-group differences in hyper-fibrinolysis, thromboembolic complications, and postoperative seizures.

Researchers hypothesized that goal-directed TXA administration using viscoelastic field tests would not be inferior to the empirical TXA administration strategy in reducing postoperative bleeding and hyper-fibrinolysis. Researchers also expect that goal-directed TXA administration would be beneficial in lowering TXA-induced thromboembolic complications and seizure risks.

ELIGIBILITY:
Inclusion Criteria:

* patients who will undergo elective cardiovascular surgery employing cardiopulmonary bypass
* patients who provide written informed consent

Exclusion Criteria:

* pregnancy
* refusal of allogenic blood transfusion
* taking thrombin
* history of thromboembolic and familial hypercoagulability disease
* recent history of myocardial infarction or ischemic cerebral infarction (within 90 days)
* hypersensitive to TXA
* histroy of convulsion or epilepsy
* taking hemodialysis
* history of Heparin-induced thrombocytopenia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 764 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
postoperative bleeding | 24 hours
  bleeding amount though chest drainage tubes during the 1st postoperative 24 hour

SECONDARY OUTCOMES:
postoperative transfusion amount | 24 hours
  amounts of transfused red blood cells, plasma, platelet and cryoprecipitate
postoperative transfusion rate | 24 hours
  incidents of red blood cells, plasma, platelet and cryoprecipitate transfusions
the lowest postoperative hemoglobin value | 24 hours
  the nadir hemoglobin value during one postoperative days
incidence of reoperation | 1 week
  incidence of reoperation due to postoperative bleeding
amount of intraoperative cell salvage | 1 hour
  amounts of infused salvaged blood
viscoelastic whole blood profile | 1 hour
  values of intraoperative CT-EXTEM, CFT-EXTEM, A10-EXTEM, MCF-EXTEM, ML-EXTEM, CT-FIBTEM, CFT-FIBTEM, A10-FIBTEM, MCF-FIBTEM, ML-FIBTEM in rotational thromboelastometry
incidence of seizure | 1 week
  incidence of postoperative seizure till the hospital discharge
incidence of thromboembolic complications | 1 week
  incidence of postoperative myocardia infarction, stroke, pulmonary embolism, gut infarction till the hospital discharge
duration of mechanical ventilation | 1 week
  duration of postoperative ventilatory care
length of stays in the ICU and hospital | 1 week
  duration of stay in the ICU and hospital
total cost | 2 week
  total expense paid at the discharge
incidence of taking renal replacement therapy | 1 week
  incidence of taking hemodylaysis
incidence of acute kidney injury | 1 week
  diagnosed by KIDGO criteria
incidence of postoperative delirium | 1 week
  delirium digested by CAM-ICU
incidence of applying for mechanical circulatory support | 1 week
  incidences of applying IABP, ECMO, VAD
in-hospital mortality | 1 week
  hospital death
central laboratory blood tests | 1 week
  hemoglobin, platelet number, Prothrombin timeI activated partial thromboplastin timePTT , fibrinogen concentration, d-dimer

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD, PhD, Principal Investigator — Konkuk University Medical Center
Locations (3):
- South Korea (3):
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nam JS, Oh CS, Kim JY, Choi DK, Oh AR, Park J, Lee JH, Yun SC, Kim KW, Jang MU, Kim TY, Choi IC. A multi-center, double-blind, placebo-controlled, randomized, parallel-group, non-inferiority study to compare the efficacy of goal-directed tranexamic acid administration based on viscoelastic test versus preemptive tranexamic acid administration on postoperative bleeding in cardiovascular surgery (GDT trial). Trials. 2024 Sep 27;25(1):623. doi: 10.1186/s13063-024-08467-1. PMID 39334224